CLINICAL TRIAL: NCT04202679
Title: A Randomized, Double Blind, Placebo-controlled, Multi-center, Parallel Group Study to Evaluate the Efficacy and Safety of Dupilumab in Patients With Prurigo Nodularis Who Are Inadequately Controlled on Topical Prescription Therapies or When Those Therapies Are Not Advisable
Brief Title: Study of Dupilumab for the Treatment of Patients With Prurigo Nodularis, Inadequately Controlled on Topical Prescription Therapies or When Those Therapies Are Not Advisable (PRIME2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16460; 2019-003801-90; U1111-1241-8174 (Other: UTN)
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Neurodermatitis
MeSH Terms: conditions — Neurodermatitis | interventions — dupilumab; Calcineurin Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matched to dupilumab 600 milligrams (mg) (loading dose), subcutaneously (SC) on Day 1 followed by placebo matched to dupilumab 300 mg once every 2 weeks (q2w) for 24 weeks added to background therapy of topical corticosteroids/topical calcineurin inhibitors (TCS/TCI) at stable dose.
  Interventions: Drug: Placebo; Drug: Moisturizers; Drug: Low to medium potent topical corticosteroids; Drug: Topical calcineurin inhibitors
- Dupilumab 300 mg Q2W (Experimental): Participants received dupilumab at a loading dose of 600 mg, SC on Day 1 followed by dupilumab 300 mg q2w for 24 weeks added to background therapy of TCS/TCI at stable dose.
  Interventions: Drug: Dupilumab SAR231893; Drug: Moisturizers; Drug: Low to medium potent topical corticosteroids; Drug: Topical calcineurin inhibitors

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Dupilumab 300 mg Q2W
Drug: Placebo — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Placebo
Drug: Moisturizers — Pharmaceutical form:
  Route of administration: Topical
Drug: Low to medium potent topical corticosteroids — Pharmaceutical form:
  Route of administration: Topical
Drug: Topical calcineurin inhibitors — Pharmaceutical form:
  Route of administration: Topical

SUMMARY:
Primary Objective:

To demonstrate the efficacy of dupilumab on itch response in participants with prurigo nodularis (PN), inadequately controlled on topical prescription therapy or when those therapies are not advisable.

Secondary Objectives:

To demonstrate the efficacy of dupilumab on additional itch endpoints in participants with PN, inadequately controlled on topical prescription therapy or when those therapies are not advisable.

To demonstrate efficacy of dupilumab on skin lesions of PN. To demonstrate the improvement in health-related quality of life. To evaluate safety outcome measures. To evaluate immunogenicity of dupilumab.

DETAILED DESCRIPTION:
The duration of study for each participant included 2-4 weeks of screening period, 24 weeks of treatment period and 12 weeks of post treatment period.

ELIGIBILITY:
Inclusion criteria :

Must be 18 to 80 years of age, at the time of signing the informed consent.

With a clinical diagnosis of PN defined by all of the following:

* Diagnosed by a dermatologist for at least 3 months before the Screening visit.
* On the Worst Itch Numeric Rating Scale (WI-NRS) ranging from 0 to 10, participants must have an average worst itch score of >=7 in the 7 days prior to Day1.
* Participants must have a minimum of 20 PN lesions in total on both legs, and/or both arms and/or trunk, at Screening visit and Day 1
* History of failing a 2-week course of medium-to-superpotent topical corticosteroids (TCS) or when TCS are not medically advisable
* Have applied a stable dose of topical emollient (moisturizer) once or twice daily for at least 5 out of the 7 consecutive days immediately before Day 1.

Must be willing and able to complete a daily symptom eDiary for the duration of the study.

Exclusion criteria:

Participants were excluded from the study if any of the following criteria apply:

* Presence of skin morbidities other than PN and mild atopic dermatitis that may interfere with the assessment of the study outcomes.
* PN secondary to medications.
* PN secondary to medical conditions such as neuropathy or psychiatric disease.
* Within 6 months before the screening visit, or documented diagnosis of moderate to severe atopic dermatitis from screening visit to randomization visit.
* Severe concomitant illness(es) under poor control that, in the investigator's judgment, would adversely affect the participant's participation in the study.
* Severe renal conditions (eg, participants with uremia and/or on dialysis).
* Participants with uncontrolled thyroid disease.
* Active tuberculosis or non-tuberculous mycobacterial infection, or a history of incompletely treated tuberculosis unless documented adequately treated.
* Diagnosed active endoparasitic infections; suspected or high risk of endoparasitic infection, unless clinical and (if necessary) laboratory assessment have ruled out active infection before randomization.
* Active chronic or acute infection (except HIV) requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals within 2 weeks before the screening visit and during the screening period.
* Known or suspected immunodeficiency.
* Active malignancy or history of malignancy within 5 years before the Baseline visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (57):
- United States (7):
  - Investigational Site Number :8400054, Fort Smith, Arkansas
  - Investigational Site Number :8400008, Sacramento, California
  - Investigational Site Number :8400005, Pembroke Pines, Florida
  - Investigational Site Number :8400002, Plainfield, Indiana
  - Investigational Site Number :8400003, Baltimore, Maryland
  - Investigational Site Number :8400006, East Windsor, New Jersey
  - Investigational Site Number :8400001, Sugar Land, Texas
- Canada (6):
  - Investigational Site Number :1240002, Calgary, Alberta
  - Investigational Site Number :1240006, Surrey, British Columbia
  - Investigational Site Number :1240007, Markham, Ontario
  - Investigational Site Number :1240008, Newmarket, Ontario
  - Investigational Site Number :1240001, Toronto, Ontario
  - Investigational Site Number :1240009, Saskatoon, Saskatchewan
- Chile (6):
  - Investigational Site Number :1520005, Valdivia, Los Ríos Region
  - Investigational Site Number :1520006, Osorno, Reg Metropolitana de Santiago
  - Investigational Site Number :1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number :1520002, Santiago
- France (8):
  - Investigational Site Number :2500007, Bordeaux
  - Investigational Site Number :2500001, Brest
  - Investigational Site Number :2500008, Le Mans
  - Investigational Site Number :2500002, Lille
  - Investigational Site Number :2500006, Lyon
  - Investigational Site Number :2500004, Paris
  - Investigational Site Number :2500005, Reims
  - Investigational Site Number :2500003, Toulouse
- Hungary (4):
  - Investigational Site Number :3480004, Debrecen
  - Investigational Site Number :3480002, Orosháza
  - Investigational Site Number :3480005, Pécs
  - Investigational Site Number :3480003, Szeged
- Italy (4):
  - Investigational Site Number :3800001, Rozzano, Milano
  - Investigational Site Number :3800004, Ancona
  - Investigational Site Number :3800003, Catanzaro
  - Investigational Site Number :3800002, Milan
- Portugal (3):
  - Investigational Site Number :6200001, Coimbra
  - Investigational Site Number :6200002, Lisbon
  - Investigational Site Number :6200003, Porto
- South Korea (6):
  - Investigational Site Number :4100002, Busan, Busan
  - Investigational Site Number :4100003, Bucheon-si, Gyeonggi-do
  - Investigational Site Number :4100007, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number :4100005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100006, Seoul, Seoul-teukbyeolsi
- Spain (7):
  - Investigational Site Number :7240009, Badalona, Barcelona [Barcelona]
  - Investigational Site Number :7240001, Pontevedra, Galicia [Galicia]
  - Investigational Site Number :7240008, Santullano, Principality of Asturias
  - Investigational Site Number :7240004, Córdoba
  - Investigational Site Number :7240007, Madrid
  - Investigational Site Number :7240003, Valencia
  - Investigational Site Number :7240002, Zaragoza
- Taiwan (5):
  - Investigational Site Number :1580005, Hsinchu
  - Investigational Site Number :1580006, Kaohsiung City
  - Investigational Site Number :1580008, Taichung
  - Investigational Site Number :1580001, Taipei
  - Investigational Site Number :1580002, Taipei
- Investigational Site Number :8260001, Redhill, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Yosipovitch G, Kim BS, Koo JY, Chen Z, Wiggins S, Zahn J, Sugerman P, Haddad EB, Cyr SL. Dupilumab Reduces Pruritus in Clinically Distinct Dermatologic Diseases: Data from Clinical Trials on Atopic Dermatitis, Prurigo Nodularis, and Chronic Spontaneous Urticaria. Dermatol Ther (Heidelb). 2025 Nov 22. doi: 10.1007/s13555-025-01596-8. Online ahead of print. PMID 41272364
- [Derived] Kim BS, Goncalo M, Ugajin T, Gao XH, Praestgaard AH, Makhija M, Zahn J, Bansal A, Wiggins S. Efficacy and Safety of Dupilumab in Adults with Prurigo Nodularis with or Without Atopic Comorbidities: A Subgroup Analysis from Two Randomized Phase III Clinical Trials. Am J Clin Dermatol. 2026 Jan;27(1):167-180. doi: 10.1007/s40257-025-00993-1. Epub 2025 Nov 11. PMID 41219577
- [Derived] Kwatra SG, Yosipovitch G, Kim B, Stander S, Rhoten S, Ivanescu C, Haeusler N, Brookes E, Msihid J, Makhija M, Bansal A, Thomas RB, Bahloul D. Worst Itch Numeric Rating Scale for Prurigo Nodularis: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Dermatol. 2024 Aug 1;160(8):813-821. doi: 10.1001/jamadermatol.2024.1634. PMID 38865146
- [Derived] Yosipovitch G, Mollanazar N, Stander S, Kwatra SG, Kim BS, Laws E, Mannent LP, Amin N, Akinlade B, Staudinger HW, Patel N, Yancopoulos GD, Weinreich DM, Wang S, Shi G, Bansal A, O'Malley JT. Dupilumab in patients with prurigo nodularis: two randomized, double-blind, placebo-controlled phase 3 trials. Nat Med. 2023 May;29(5):1180-1190. doi: 10.1038/s41591-023-02320-9. Epub 2023 May 4. PMID 37142763
- See also: EFC16460 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25247&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 57 sites in 11 countries. A total of 221 participants were screened from 16 January 2020 to 24 February 2021, out of which 61 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 160 participants were randomized in 1:1 ratio to receive study interventions (placebo or dupilumab) by interactive response technology (IRT).
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Started | 82 | 78
Treated | 82 | 77
Completed | 56 | 72
Not Completed | 26 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Poor compliance to protocol | 1 | 0
Not completed — Withdrawal by Subject | 23 | 6

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Placebo: Participants received placebo matched to dupilumab 600 mg (loading dose), SC on Day 1 followed by placebo matched to dupilumab 300 mg q2w for 24 weeks added to background therapy TCS/TCI at stable dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg Q2W | Total
Number analyzed (Participants) | 82 | 78 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (15.2) | 51.0 (15.8) | 48.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 31 | 26 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 27 | 25 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 48 | 48 | 96
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 4 Points Improvement (Reduction) From Baseline in Worst-Itch Numeric Rating Scale (WI-NRS) Scores at Week 12
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity. Percentage of participants with >=4 points improvement (reduction) from baseline in WI-NRS scores at Week 12 is reported in this outcome measure.
Time Frame: Baseline, Week 12
Population: Analysis was performed on intent-to-treat (ITT) population which included all participants with a treatment kit number allocated and recorded in the IRT database analyzed according to the treatment group allocated by randomization regardless of if treatment kit was used or not.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo matched to dupilumab 600 mg (loading dose), SC on Day 1 followed by placebo matched to dupilumab 300 mg q2w for 24 weeks added to background therapy of TCS/TCI at stable dose.
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants | 22.0 | 37.2
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when primary outcome measure was statistically significant at two-sided 0.05; Test type: Superiority; p = 0.0216, Cochran-Mantel-Haenszel — Threshold of significance at 0.05 level; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.08 to 5.00] — Dupilumab 300 mg q2w versus Placebo

2. Secondary Outcome: Percentage of Participants With >=4 Points Improvement (Reduction) From Baseline in WI-NRS Scores at Week 24
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity. Percentage of participants with >=4 points improvement (reduction) from baseline in WI-NRS scores at Week 24 is reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants | 19.5 | 57.7
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at two-sided 0.05; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold of significance at 0.05 level; Odds Ratio (OR) = 9.0, 95% CI 2-sided [3.56 to 22.66] — Dupilumab 300 mg q2w versus Placebo

3. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment For Prurigo Nodularis-Stage (IGA PN-S) Scores of 0 or 1 at Week 24
Description: IGA PN-S is an instrument used to assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe prurigo nodularis. In this outcome measure, percentage of participants with IGA PN-S score of either 0 (clear) or 1 (almost clear) has been reported.
Time Frame: At Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants | 15.9 | 44.9
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold of significance at 0.05 level; Odds Ratio (OR) = 4.4, 95% CI 2-sided [2.02 to 9.55] — Dupilumab 300 mg q2w versus Placebo

4. Secondary Outcome: Percentage of Participants With Both an Improvement (Reduction) in WI-NRS by >=4 Points and an IGA PN-S Score of 0 or 1 From Baseline at Week 24
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch), higher scores indicated more severity. IGA PN-S assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4 where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicated greater severity. Percentage of participants with both an improvement (reduction) in WI-NRS by >=4 Points (from Baseline) and an IGA PN-S score of 0 or 1 were reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants | 8.5 | 32.1
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — Threshold of significance at 0.05 level; Odds Ratio (OR) = 6.1, 95% CI 2-sided [2.03 to 18.11] — Dupilumab 300 mg q2w versus Placebo

5. Secondary Outcome: Percentage of Participants With IGA PN-S Scores of 0 or 1 at Week 12
Description: as for outcome 3
Time Frame: At Week 12
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants | 12.2 | 25.6
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0194, Cochran-Mantel-Haenszel — Threshold of significance at 0.05 level; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.13 to 7.52] — Dupilumab 300 mg q2w versus Placebo

6. Secondary Outcome: Percent Change From Baseline in WI-NRS Scores at Week 24
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity. Least squares (LS) means and standard error (SE) were obtained from Analysis of covariance (ANCOVA) model.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 74 | 76
percent change | -36.18 (6.21) | -59.34 (6.39)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold of significance at 0.05 level; LS mean difference = -23.16, 95% CI 2-sided [-33.81 to -12.51] — Dupilumab 300 mg q2w versus Placebo

7. Secondary Outcome: Change From Baseline in Health-related Quality of Life (HRQoL) as Measured by Dermatology Life Quality Index (DLQI) at Week 24
Description: DLQI is developed to measure dermatology specific HRQoL in adult participants. It comprises of set of 10 questions assessing the impact of skin disease on participants' HRQoL over the previous week. Responses to each question were assessed on a 4-point Likert scale ranged from 0 (not at all) to 3 (very much). Scores from all 10 questions added up to give total DLQI scores ranged from 0 (not at all) to 30 (very much), higher scores indicated more impact on quality of life. LS means and SE were obtained from ANCOVA model.
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 75 | 77
score on a scale | -6.77 (1.18) | -13.16 (1.21)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold of significance at 0.05 level; LS mean difference = -6.39, 95% CI 2-sided [-8.42 to -4.36] — Dupilumab 300 mg q2w versus Placebo

8. Secondary Outcome: Change From Baseline in Skin Pain-NRS at Week 24
Description: Skin Pain-NRS was used to measure skin pain intensity. Participants were asked daily to rate the intensity of their worst skin pain over the past 24 hours, using a 11-point scale ranging from 0 ("No pain") to 10 ("Worst possible pain"). Higher scores indicated more severity. LS means and SE were obtained from ANCOVA model.
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 74 | 76
score on a scale | -2.74 (0.51) | -4.35 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA — Threshold of significance at 0.05 level; LS mean difference = -1.61, 95% CI 2-sided [-2.49 to -0.73] — Dupilumab 300 mg q2w versus Placebo

9. Secondary Outcome: Change From Baseline in Sleep-NRS at Week 24
Description: Sleep-NRS was used to measure sleep intensity. Participants were asked to rate their sleep quality on their past night upon awakening, using a 11-point NRS ranging from 0 to 10, where 0 = worst possible sleep and 10 = best possible sleep. Higher scores indicated less severity. LS means and SE were obtained from ANCOVA model.
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 74 | 76
score on a scale | 0.76 (0.45) | 1.30 (0.46)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1658, ANCOVA — Threshold of significance at 0.05 level; LS mean difference = 0.54, 95% CI 2-sided [-0.22 to 1.30] — Dupilumab 300 mg q2w versus Placebo

10. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Total Score at Week 24
Description: HADS is a 14-item self-administered questionnaire that consists of 2 scales, one measuring anxiety (HADS-A), and the other measuring depression (HADS-D). Each subscale comprised of 7 items with a scoring range from 0 (less severity of anxiety and depression) to 21 (greater severity of anxiety and depression symptoms) for each subscale. The total HADS score ranges from 0 (less severity) to 42 (more severity), with a high score indicative of a severe anxiety and/or depression level. LS means and SE were obtained from ANCOVA model.
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 76 | 77
score on a scale | -2.59 (1.03) | -5.55 (1.06)

11. Secondary Outcome: Probability of Participants With an Improvement (Reduction) in WI-NRS by >=4 From Baseline at Week 24
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity. Probability of participants with an improvement (reduction) in WI-NRS at Week 24 was based on Kaplan-Meier estimates and was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population.
Measure: Number (95% Confidence Interval); unit: probability of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
probability of participants | 0.353 [0.250 to 0.457] | 0.670 [0.552 to 0.764]

12. Secondary Outcome: Change From Baseline in WI-NRS Scores at Weeks 12 and 24
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity. LS means and SE were obtained from ANCOVA model.
Time Frame: Baseline, Weeks 12 and 24
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 79 | 77
score on a scale
  Week 12 | -3.04 (0.46) | -4.11 (0.47)
  Week 24: number analyzed (Participants) | 74 | 76
  Week 24 | -3.10 (0.53) | -5.05 (0.54)

13. Secondary Outcome: Percent Change From Baseline in WI-NRS Scores at Weeks 2, 4 and 12
Description: as for outcome 12
Time Frame: Baseline, Weeks 2, 4 and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 81 | 77
percent change
  Week 2 | -15.61 (3.06) | -17.41 (3.15)
  Week 4 | -22.61 (4.00) | -30.09 (4.12)
  Week 12: number analyzed (Participants) | 79 | 77
  Week 12 | -35.83 (5.42) | -48.86 (5.59)

14. Secondary Outcome: Percent Change From Baseline in WI-NRS Scores at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24
Description: as for outcome 12
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24
Population: Analysis was performed on ITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percent change
  Week 1 | -9.49 (2.12) | -8.66 (2.18)
  Week 2: number analyzed (Participants) | 81 | 77
  Week 2 | -15.61 (3.06) | -17.41 (3.15)
  Week 3: number analyzed (Participants) | 81 | 77
  Week 3 | -20.44 (3.66) | -25.26 (3.77)
  Week 4: number analyzed (Participants) | 81 | 77
  Week 4 | -22.61 (4.00) | -30.09 (4.12)
  Week 5: number analyzed (Participants) | 81 | 77
  Week 5 | -25.21 (4.21) | -34.41 (4.33)
  Week 6: number analyzed (Participants) | 80 | 77
  Week 6 | -27.87 (4.33) | -36.98 (4.46)
  Week 7: number analyzed (Participants) | 78 | 76
  Week 7 | -28.99 (4.69) | -39.30 (4.84)
  Week 8: number analyzed (Participants) | 79 | 77
  Week 8 | -30.45 (4.56) | -41.32 (4.70)
  Week 9: number analyzed (Participants) | 79 | 77
  Week 9 | -34.86 (4.89) | -47.08 (5.04)
  Week 10: number analyzed (Participants) | 78 | 76
  Week 10 | -32.90 (5.04) | -44.65 (5.20)
  Week 11: number analyzed (Participants) | 79 | 77
  Week 11 | -34.64 (5.25) | -45.98 (5.41)
  Week 12: number analyzed (Participants) | 79 | 77
  Week 12 | -35.83 (5.42) | -48.86 (5.59)
  Week 13: number analyzed (Participants) | 79 | 77
  Week 13 | -34.49 (5.69) | -48.32 (5.86)
  Week 14: number analyzed (Participants) | 79 | 77
  Week 14 | -36.60 (5.71) | -50.67 (5.88)
  Week 15: number analyzed (Participants) | 79 | 77
  Week 15 | -35.96 (5.74) | -51.89 (5.91)
  Week 16: number analyzed (Participants) | 77 | 77
  Week 16 | -37.80 (5.74) | -54.36 (5.91)
  Week 17: number analyzed (Participants) | 77 | 77
  Week 17 | -39.15 (5.98) | -55.95 (6.15)
  Week 18: number analyzed (Participants) | 77 | 77
  Week 18 | -40.38 (6.15) | -56.80 (6.32)
  Week 19: number analyzed (Participants) | 76 | 77
  Week 19 | -40.03 (6.05) | -57.75 (6.23)
  Week 20: number analyzed (Participants) | 74 | 77
  Week 20 | -36.12 (5.94) | -56.80 (6.10)
  Week 21: number analyzed (Participants) | 74 | 76
  Week 21 | -36.43 (6.16) | -56.91 (6.34)
  Week 22: number analyzed (Participants) | 74 | 76
  Week 22 | -37.34 (6.19) | -58.78 (6.33)
  Week 23: number analyzed (Participants) | 73 | 75
  Week 23 | -36.87 (6.19) | -59.43 (6.32)
  Week 24: number analyzed (Participants) | 74 | 76
  Week 24 | -36.18 (6.21) | -59.34 (6.39)

15. Secondary Outcome: Percentage of Participants With Improvement (Reduction) in WI-NRS >=4 Points From Baseline at Week 4
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity. Percentage of participants with improvement (Reduction) in WI-NRS scale by >=4 Points at Week 4 is reported in this outcome measure.
Time Frame: Baseline, Week 4
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants | 7.3 | 16.7

16. Secondary Outcome: Percentage of Participants Achieving >=4 Points Improvement (Reduction) From Baseline in WI-NRS Scores at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24
Description: WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated more severity. Percentage of participants achieving >=4 points improvement (reduction) from Baseline in WI-NRS scores at Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24 is reported in this outcome measure.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants
  Week 1 | 1.2 | 1.3
  Week 2 | 1.2 | 5.1
  Week 3 | 6.1 | 12.8
  Week 4 | 7.3 | 16.7
  Week 5 | 4.9 | 17.9
  Week 6 | 13.4 | 23.1
  Week 7 | 15.9 | 24.4
  Week 8 | 14.6 | 28.2
  Week 9 | 24.4 | 32.1
  Week 10 | 18.3 | 32.1
  Week 11 | 17.1 | 33.3
  Week 12 | 22.0 | 37.2
  Week 13 | 19.5 | 39.7
  Week 14 | 22.0 | 39.7
  Week 15 | 20.7 | 44.9
  Week 16 | 19.5 | 44.9
  Week 17 | 23.2 | 47.4
  Week 18 | 24.4 | 48.7
  Week 19 | 23.2 | 51.3
  Week 20 | 20.7 | 51.3
  Week 21 | 20.7 | 48.7
  Week 22 | 22.0 | 50.0
  Week 23 | 20.7 | 55.1
  Week 24 | 19.5 | 57.7

17. Secondary Outcome: Onset of Action Based on Change From Baseline in WI-NRS at Week 4
Description: Onset of action was defined as the first p<0.05 difference from placebo in the weekly average WI-NRS that remained significant at subsequent measurements. WI-NRS is a validated measure of itch severity. Participants were asked daily to rate the intensity of their worst pruritus (itch) over the past 24 hours, using a 11-point scale ranging from 0 (no itch) to 10 (worst imaginable itch). Higher scores indicated greater severity.
Time Frame: Baseline, Week 4
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 81 | 77
score on a scale | -1.94 (0.33) | -2.55 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg Q2W; Test type: Superiority; p = 0.0370, ANCOVA — Threshold of significance was <0.05; LS mean difference = -0.61, 95% CI 2-sided [-1.18 to -0.04] — Dupilumab 300 mg q2w versus Placebo

18. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment for PN-Stage (IGA PN-S) Score of 0 or 1 at Weeks 4 and 8
Description: IGA PN-S is an instrument used to assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4: where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe prurigo nodularis. In this outcome measure, percentage of participants with IGA PN-S score of either 0 (clear) or 1 (almost clear) has been reported.
Time Frame: At Weeks 4 and 8
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants
  Week 4 | 6.1 | 7.7
  Week 8 | 9.8 | 15.4

19. Secondary Outcome: Change From Baseline in IGA PN-S Scores at Weeks 4, 8, 12, and 24
Description: IGA PN-S is an instrument used to assess the overall number and thickness of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4: where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. Higher scores indicate severe prurigo nodularis. LS means and SE were obtained from ANCOVA model.
Time Frame: Baseline, Weeks 4, 8, 12, and 24
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 80 | 77
score on a scale
  Week 4 | -0.54 (0.13) | -0.69 (0.13)
  Week 8: number analyzed (Participants) | 76 | 76
  Week 8 | -0.79 (0.17) | -1.19 (0.17)
  Week 12: number analyzed (Participants) | 78 | 77
  Week 12 | -0.86 (0.18) | -1.47 (0.18)
  Week 24: number analyzed (Participants) | 74 | 77
  Week 24 | -1.07 (0.20) | -2.03 (0.20)

20. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment for PN-Activity (IGA PN-A) Score of 0 or 1 at Weeks 4, 8, 12 and 24
Description: The IGA PN-A is an instrument used to assess the overall activity of PN lesions at a given time point, as determined by the investigator. It consists of a 5-point scale ranging from 0 to 4: where 0 = clear (0% nodules showing excoriations/crusts), 1 = almost clear (up to 10% nodules showing excoriations/crusts), 2 = mild (11-25% nodules showing excoriations/crusts), 3 = moderate (26-75% nodules showing excoriations/crusts) and 4 = severe (76-100% of nodules showing excoriations/crusts). Higher scores indicate severe prurigo nodularis. In this outcome measure, percentage of participants with IGA PN-A score of either 0 (clear) or 1 (almost clear) has been reported.
Time Frame: At Weeks 4, 8, 12 and 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 78
percentage of participants
  Week 4 | 4.9 | 14.1
  Week 8 | 15.9 | 23.1
  Week 12 | 19.5 | 42.3
  Week 24 | 18.3 | 51.3

21. Secondary Outcome: Change From Baseline in HRQoL, as Measured by DLQI at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 78 | 77
score on a scale | -7.05 (1.12) | -12.07 (1.16)

22. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the treatment-emergent (TE) period (time from the first investigational medicinal product [IMP] administration to the last IMP administration + 14 weeks).
Time Frame: From the first IMP administration to the last IMP administration + 14 weeks (i.e., up to 36 weeks)
Population: Analysis was performed on safety population which included all participants who received at least 1 dose of study intervention analyzed according to the intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 82 | 77
Participants
  TEAEs | 47 | 47
  TESAEs | 4 | 2

23. Secondary Outcome: Number of Participants With Treatment-emergent and Treatment Boosted Antidrug Antibodies (ADA)
Description: ADA response was categorized as: Treatment emergent and Treatment-boosted. Treatment emergent ADAs were defined as a participant with no positive assay response at baseline but with a positive assay response during the entire TEAE period. Treatment boosted ADAs: defined as participants with a positive ADA assay response at baseline and with at least a 4-fold increase in titer compared to baseline during the TE period (time from the first IMP administration to the last IMP administration + 14 weeks). Titer values were defined as low titer (< 1,000); moderate (1,000 <= titer <= 10,000) and high titer (> 10,000).
Time Frame: From the first IMP administration to the last IMP administration + 14 weeks (i.e., up to 36 weeks)
Population: Analysis was performed on ADA population which included all participants who received at least one dose of the study drug and had at least one non-missing ADA result after first dose of study drug. Participants were analyzed according to the intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 80 | 76
Participants
  Treatment-emergent ADAs | 1 | 7
  Treatment-boosted ADAs | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first IMP administration to the last IMP administration + 14 weeks (i.e., up to 36 weeks)
Description: Reported AEs were TEAEs that developed/worsened in grade or became serious during TE period (defined as the time from the first IMP administration to the last IMP administration + 14 weeks). Analysis was performed on safety population.
Arm/Group | Placebo | Dupilumab 300 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/77
Serious Adverse Events (participants affected / at risk) | 4/82 | 2/77
Other Adverse Events (participants affected / at risk) | 10/82 | 11/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Dupilumab 300 mg Q2W (N=77)
Pelvic Inflammatory Disease (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1)
Cutaneous T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large Granular Lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cauda Equina Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | Dupilumab 300 mg Q2W (N=77)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 5 (9) | 4 (4)
Accidental Overdose (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT04202679/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04202679/SAP_001.pdf